CLINICAL TRIAL: NCT02487862
Title: Evaluating the Adjunctive Effect of Stress Reduction Protocol in the Non-Surgical Periodontal Therapy of Chronic Periodontitis Subjects Associated With Stress: A Randomized Control Pilot Study
Brief Title: Role of Stress Reduction Protocol on Outcome of Periodontal Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KCDS
Record Dates: First submitted 2015-05-12; First posted 2015-07-02 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-09

CONDITIONS: Combat and Operational Stress Reaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Screening (No Intervention): Participants were screened for the inclusion and exclusion criteria to select the study group. No intervention has been done.
- catagerizing the study population (Placebo Comparator): The selected participants where assigned into respective groups
  Interventions: Behavioral: Stress Reduction Protocol
- Stress Reduction Protocol (No Intervention): Participants were evaluated for the outcome of the intervention.

INTERVENTIONS:
Behavioral: Stress Reduction Protocol — Stress Reduction Protocol
  Arms: catagerizing the study population

SUMMARY:
Psychological conditions, particularly psychosocial stress, have been implicated as risk indicators for periodontal disease. Minimal evidence in literature exists to assess the effect of stress reduction therapy (SRT) in the outcome of non-surgical periodontal therapy (NSPT). Hence, the present study was aimed at exploring the possibility of employing SRT in stressed subjects (assessed using questionnaire data and serum cortisol level) as an adjunctive intervention in the management of periodontal diseases.

DETAILED DESCRIPTION:
Periodontitis is a multifactorial disease where microbial dental biofilms are considered to be a key etiological agent for the initiation & progression of the inflammatory process. Apart from the microbial biofilms, several other risk factors have been associated with increased susceptibility, progression and severity of periodontal diseases such as systemic diseases, genetic polymorphisms, socio-economic or educational status, tobacco smoking, oral hygiene level and psychological stress.

With respect to other possible factors influencing chronic periodontitis, more direct evidence has emerged that stress, depression and anxiety contribute to the development of periodontitis in odds ratio of 1:2. Further, it has been shown that subjects with stress are more prone to develop periodontal disease than subjects without stress. It is speculated that chronic stress contribute to the development of periodontitis by having a net negative effect on the immunological response of body or by health related risk behaviors such as smoking, over eating and lessen compliance with the preventive behavior or even both. In addition, it has been found that patients experiencing stress were slower in recovery from periodontal treatment compared to subjects who are not experiencing stress.

Interestingly, the impact of stress on the pathogenesis and periodontal treatment outcomes depends upon the individuals coping ability. Literature evidence shows that emotional-focused coping individuals (defensive coping, resigned coping, distractive coping which are advantageous in the short term) have more advanced disease and poor response to non-surgical periodontal treatment when compared to problem focused coping (i.e. active coping). Hence, assessment of a patient's stress level, their coping ability and stress management might be of value in understanding psychological effects on periodontal health and its disease process, which will be helpful in future preventive care. Considering these facts, we hypothesize that if stress is causally related to the worsening of parameters in a chronic periodontitis patient, its alleviation might result in an additive response to the conventional periodontal therapy. However, till date, there are no intervention studies on possibility of employing psychological intervention (stress reduction therapy) as adjunctive measure in the treatment of periodontitis subjects with unfavorable psychological background. Hence, considering this hypothesis, the present study is conducted which is first of its kind, to explore and evaluate, if intervention focused on stress management enhancement training may serve as adjunctive role in non-surgical treatment of periodontal diseases by monitoring the improvements in periodontal condition through clinical parameters and correlating with stress marker like salivary cortisol levels and Derogatis stress profile (DSP) scores.

ELIGIBILITY:
Inclusion Criteria:

* patients within the age group of 30 to 55 years,
* systemically healthy stressed & unstressed individuals with chronic periodontitis and
* who were co-operative and willing to attend follow up visits

Exclusion Criteria:

* patients on corticosteroids and antipsychotic drug therapy,
* who had received any periodontal therapy,
* surgical or non- surgical within the past six months of baseline examination,
* Smokers,
* no prior history of non-surgical periodontal therapy within 6 months,
* with less than 20 permanent teeth remaining,
* history of psychiatric treatment within past 6 months,
* known systemic diseases and conditions.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan BV, MDS, Study Director — Krishnadevaraya College of Dental Sciences
Locations (1):
- Krishnadevaraya College of dental sciences, Banglore, Karnataka, India

REFERENCES:
- [Result] Kiecolt-Glaser JK, Preacher KJ, MacCallum RC, Atkinson C, Malarkey WB, Glaser R. Chronic stress and age-related increases in the proinflammatory cytokine IL-6. Proc Natl Acad Sci U S A. 2003 Jul 22;100(15):9090-5. doi: 10.1073/pnas.1531903100. Epub 2003 Jul 2. PMID 12840146
- See also: Reference Article — http://www.ncbi.nlm.nih.gov/pubmed/12840146